CLINICAL TRIAL: NCT02412449
Title: A Randomized, Open-Label, Single-Dose, Three-Period Crossover Study in Healthy Adults to Assess the Relative Bioavailability of Test and Reference Formulations of AKB-6548 Tablets and to Evaluate the Effect of Food on the Bioavailability of AKB-6548
Brief Title: Relative Bioavailability of Two Formulations of AKB-6548 and the Food Effect of a New Tablet in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AKB-6548-CI-0013
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Anemia; Chronic kidney disease; CKD; Renal impairment; Chronic renal insufficiency; Ferrous sulfate; Iron; End stage renal disease; Dialysis; Oral anemia treatment; Bioavailability; Erythropoietin; Hypoxia-inducible factor; Volunteers
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency; Kidney Failure, Chronic | interventions — vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): AKB-6548
  Interventions: Drug: AKB-6548 tablet, reference formulation given in the fasted state
- Treatment B (Experimental): AKB-6548
  Interventions: Drug: AKB-6548 tablet, test formulation given in the fasted state.
- Treatment C (Experimental): AKB-6548
  Interventions: Drug: AKB-6548 tablet, test formulation given in the fed state

INTERVENTIONS:
Drug: AKB-6548 tablet, reference formulation given in the fasted state
  Arms: Treatment A
Drug: AKB-6548 tablet, test formulation given in the fasted state.
  Arms: Treatment B
Drug: AKB-6548 tablet, test formulation given in the fed state
  Arms: Treatment C

SUMMARY:
The primary purpose of this study is to compare the PK parameters of a single dose of a test tablet formulation of AKB-6548 relative to a single dose of the reference AKB-6548 tablet formulation, both treatments administered without food, and to compare the PK parameters of the test tablet formulation given under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 and 55 years of age, inclusive, and with a body mass index between 18 and 30 kg/m2, inclusive.

Exclusion Criteria:

* Current or past history of cardiovascular, cerebrovascular, pulmonary, renal or liver disease.
* Positive serology results for HBsAg, HCV, and HIV at Screening.
* Significant renal impairment as evidenced by an estimated glomerular filtration rate (eGFR) of <65 mL/min
* Known active cancer (except non-melanoma skin cancer) or history of chemotherapy use within the previous 24 months.
* Current or past history of gastric or duodenal ulcers or other diseases of the GI tract (including gastric bypass surgeries) that could interfere with absorption of study drug.
* Subjects with a known history of smoking and/or have used nicotine or nicotine-containing products within the past 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Bioavailability endpoints: Area under the plasma concentration-time curve from 0 to last quantifiable concentration (AUC 0-t) of AKB-6548 | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Bioavailability endpoints: Area under the concentration time curve from time 0 to infinity (AUC 0-inf) of AKB-6548 | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Bioavailability endpoints: Maximum observed plasma concentration (Cmax) of AKB-6548 | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Food Effect Endpoint: AKB-6548 AUC 0-t for the fed versus fasted administration of AKB-6548 tablets | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Food Effect Endpoint: AKB-6548 AUC 0-inf for the fed versus fasted administration of AKB-6548 tablets | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Food Effect Endpoint: AKB-6548 Cmax for the fed versus fasted administration of AKB-6548 tablets | Multiple timepoint evaluations from pre-dose to 24 hours post-dose

SECONDARY OUTCOMES:
PK Parameters of AKB-6548: Maximum observed plasma concentration (Cmax) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK Parameters of AKB-6548: Time to reach Cmax (Tmax) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK Parameters of AKB-6548: Terminal elimination rate constant (λz) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK Parameters of AKB-6548: Terminal elimination half-life (t1/2) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK Parameters of AKB-6548: Area under the plasma concentration-time curve from 0 to last quantifiable concentration (AUC 0-t) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK Parameters of AKB-6548: AUC from time 0 to infinity (AUC 0-inf) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
AKB-6548: Apparent oral clearance (CL/F) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
AKB-6548: Apparent volume of distribution during the terminal phase (Vz/F) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (1):
- Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided